CLINICAL TRIAL: NCT04771390
Title: An Open-label, Phase I Study to Evaluate the Relative Bioavailability, Food Effect and Pharmacokinetic Linearity of 2 New Tablet Formulations (Adult and Pediatric) of Selitrectinib (BAY 2731954) in Relative to Oral Suspension and the Liquid Service Formulation in Healthy Adult Participants
Brief Title: Study to Compare How the Body Absorbs, Distributes and Excretes the Drug Selitrectinib (BAY2731954) Given as Two Different Tablet Formulations or as Liquid Formulations Including the Effect of Food on the Absorption, Distribution or Excretion of the Different Formulations in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 21416
Record Dates: First submitted 2021-02-05; First posted 2021-02-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Solid Tumors Harboring NTRK Fusion
MeSH Terms: interventions — selitrectinib; Solutions; Suspensions

STUDY DESIGN:
Intervention Model Description: Part 1: sequential and non-randomized design Part 2: cross-over and randomized design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1: Group A (Experimental): Participants will receive 3 single doses of selitrectinib in adult tablet formulation sequentially in 3 treatment periods. The washing-out period between each dose is at least 3 days
  Interventions: Drug: Selitrectinib (BAY2731954) Adult tablet
- Part 1: Group B (Experimental): Participants will receive 3 single doses of selitrectinib in pediatric tablet formulation sequentially in 3 treatment periods. The washing-out period between each dose is at least 3 days
  Interventions: Drug: Selitrectinib (BAY2731954) Pediatric tablet
- Part 2 (Group A): Dose A-B-C-D (Experimental): Participants will receive dose A, B, C and D sequentially. The washing-out period between each dose is at least 3 days
  Interventions: Drug: Selitrectinib (BAY2731954) Adult tablet; Drug: Selitrectinib (BAY2731954) Oral solution; Drug: Selitrectinib (BAY2731954) Oral suspension
- Part 2 (Group A): Dose B-C-A-D (Experimental): Participants will receive dose B, C, A and D sequentially. The washing-out period between each dose is at least 3 days
  Interventions: Drug: Selitrectinib (BAY2731954) Adult tablet; Drug: Selitrectinib (BAY2731954) Oral solution; Drug: Selitrectinib (BAY2731954) Oral suspension
- Part 2 (Group A): Dose C-A-B-D (Experimental): Participants will receive dose C, A, B and D sequentially. The washing-out period between each dose is at least 3 days
  Interventions: Drug: Selitrectinib (BAY2731954) Adult tablet; Drug: Selitrectinib (BAY2731954) Oral solution; Drug: Selitrectinib (BAY2731954) Oral suspension
- Part 2 (Group B): Dose A-B-C-D (Experimental): Participants will receive dose A, B, C and D sequentially. The washing-out period between each dose is at least 3 days
  Interventions: Drug: Selitrectinib (BAY2731954) Pediatric tablet; Drug: Selitrectinib (BAY2731954) Oral suspension
- Part 2 (Group B): Dose B-D-A-C (Experimental): Participants will receive dose B, D, A and C sequentially. The washing-out period between each dose is at least 3 days
  Interventions: Drug: Selitrectinib (BAY2731954) Pediatric tablet; Drug: Selitrectinib (BAY2731954) Oral suspension
- Part 2 (Group B): Dose C-A-D-B (Experimental): Participants will receive dose C, A, B and D sequentially. The washing-out period between each dose is at least 3 days
  Interventions: Drug: Selitrectinib (BAY2731954) Pediatric tablet; Drug: Selitrectinib (BAY2731954) Oral suspension
- Part 2 (Group B): Dose D-C-B-A (Experimental): Participants will receive dose D, C, B and A sequentially. The washing-out period between each dose is at least 3 days
  Interventions: Drug: Selitrectinib (BAY2731954) Pediatric tablet; Drug: Selitrectinib (BAY2731954) Oral suspension

INTERVENTIONS:
Drug: Selitrectinib (BAY2731954) Adult tablet — Tablet, oral administration
  Arms: Part 1: Group A; Part 2 (Group A): Dose A-B-C-D; Part 2 (Group A): Dose B-C-A-D; Part 2 (Group A): Dose C-A-B-D
Drug: Selitrectinib (BAY2731954) Pediatric tablet — Tablet, oral administration
  Arms: Part 1: Group B; Part 2 (Group B): Dose A-B-C-D; Part 2 (Group B): Dose B-D-A-C; Part 2 (Group B): Dose C-A-D-B; Part 2 (Group B): Dose D-C-B-A
Drug: Selitrectinib (BAY2731954) Oral solution — Oral solution after reconstitution
  Arms: Part 2 (Group A): Dose A-B-C-D; Part 2 (Group A): Dose B-C-A-D; Part 2 (Group A): Dose C-A-B-D
Drug: Selitrectinib (BAY2731954) Oral suspension — Oral suspension after reconstitution
  Arms: Part 2 (Group A): Dose A-B-C-D; Part 2 (Group A): Dose B-C-A-D; Part 2 (Group A): Dose C-A-B-D; Part 2 (Group B): Dose A-B-C-D; Part 2 (Group B): Dose B-D-A-C; Part 2 (Group B): Dose C-A-D-B; Part 2 (Group B): Dose D-C-B-A

SUMMARY:
In this study, the researchers will compare 2 new tablet forms of BAY2731954 with liquid oral forms of BAY2731954. A maximum of 61 healthy volunteers aged 18 to 55 will be asked to participate.

The study will have 2 parts. In part 1 researchers want to gather information how the body absorbs, distributes and excretes the drug BAY2731954 given as two different tablet formulations. Participants will take the study drugs on 3 days separated by breaks of at least 3 days between each intake. The duration of this study part will be in total of up to 6 weeks from first screening visit to follow-up visit.

In part 2 of the study researchers want to study how the body absorbs, distributes and excretes the drug BAY2731954 given as two different tablet formulations with or without food or as 2 liquid oral formulations. Participants will take the study drugs on 4 days separated by breaks of at least 3 days between each intake. The duration of the second part of study part will be in total of up to 7 weeks from first screening visit to follow-up visit.

During the study, researchers will collect blood and urine samples. In addition, doctors will check the participants' overall health. They will also ask the participants if they have any medical problems.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants who are overtly healthy as determined by the investigator or medically qualified designee based on medical evaluation including medical history, laboratory tests, physical, cardiac and neurologic examination
* Body mass index (BMI): ≥18.5 and ≤ 29.9 kg/m2, with body weight ≥50 kg
* Use of adequate contraception until 3 months after last study intervention

Key Exclusion Criteria:

* Existing relevant diseases of vital organs (e.g. liver diseases, heart diseases), central nervous system (e.g. seizures) or other organs (e.g. diabetes mellitus).
* Medical history of risk factors for Torsades de pointes (e.g. family history of Long QT Syndrome) or other arrhythmias
* Known severe allergies, allergies requiring therapy with corticosteroids, non-allergic drug reactions, or (multiple) drug allergies (excluding untreated asymptomatic seasonal allergies such as non-severe hay fever during the time of study conduct).
* Regular use of medicines
* Regular alcohol consumption
* Smoking more than 5 cigarettes daily
* History of COVID-19 or current SARS-CoV-2 infection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-07-06 (Actual)

PRIMARY OUTCOMES:
AUC | Up to 48 hours after dosing
  Area under the plasma concentration vs. time curve from 0 to infinity after single dose
  To evaluate the pharmacokinetic linearity of selitrectinib after a single dose of adult tablet and pediatric tablet and to evaluate the relative bioavailability of adult tablet and pediatric tablet formulation vs oral suspension formulation and the food effect on the bioavailability of 2 new tablet formulations
AUC(0-24) | Up to 24 hours after dosing
  Area under the plasma concentration vs. time curve from 0 to 24 hours after single dose
  To evaluate the pharmacokinetic linearity of selitrectinib after a single dose of adult tablet and pediatric tablet and to evaluate the relative bioavailability of adult tablet and pediatric tablet formulation vs oral suspension formulation and the food effect on the bioavailability of 2 new tablet formulations
Cmax | Up to 48 hours after dosing
  Maximum observed drug concentration in measured matrix after single dose administration
  To evaluate the pharmacokinetic linearity of selitrectinib after a single dose of adult tablet and pediatric tablet and to evaluate the relative bioavailability of adult tablet and pediatric tablet formulation vs oral suspension formulation and the food effect on the bioavailability of 2 new tablet formulations

SECONDARY OUTCOMES:
AUC | Up to 48 hours after dosing
  Area under the plasma concentration vs. time curve from 0 to infinity after single dose.
  To evaluate the relative bioavailability of adult tablet and pediatric tablet formulation vs oral solution
AUC(0-24) | Up to 24 hours after dosing
  Area under the plasma concentration vs. time curve from 0 to 24 hours after single dose
  To evaluate the relative bioavailability of adult tablet and pediatric tablet formulation vs oral solution
Cmax | Up to 48 hours after dosing
  Maximum observed drug concentration in measured matrix after single dose administration
  To evaluate the relative bioavailability of adult tablet and pediatric tablet formulation vs oral solution
Number of participants with treatment emergent adverse events and severity of treatment emergent adverse events | Up to 7 weeks
  Adverse events that occur or worsen after the first dose of study medication
Incidence of laboratory abnormalities, based on clinical safety laboratory assessments | Up to 7 weeks
  Hematology, clinical chemistry and urinalysis test results
Ventricular rate | Up to 7 weeks
ECG PR interval | Up to 7 weeks
ECG QT interval | Up to 7 weeks
ECG QRS duration | Up to 7 weeks
Blood pressure in mmHg | Up to 7 weeks
Heart rate in bpm | Up to 7 weeks
  bpm: beats per minute
Body temperature in Celsius | Up to 7 weeks
Respiratory rate in breaths/min | Up to 7 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Parexel International - Los Angeles, Glendale, California
  - PAREXEL International, Baltimore, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal